CLINICAL TRIAL: NCT00586079
Title: The Effect of Deep Brain Stimulation on Movement-Related Cortical Potentials in Patients With Parkinson's Disease
Brief Title: Deep Brain Stimulation in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virgilio Evidente, Professor of Neurology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-003248
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Ten patients who have had deep brain stimulation surgery for Parkinson's disease at Mayo Clinic Arizona.
  Interventions: Procedure: Deep brain stimulation surgery.
- B (Experimental): Ten patients who are scheduled to have deep brain stimulation surgery for Parkinson's disease at Mayo Clinic Arizona.
  Interventions: Procedure: Deep brain stimulation surgery.

INTERVENTIONS:
Procedure: Deep brain stimulation surgery. — Deep brain stimulation surgery.

SUMMARY:
The purpose of this study is to determine the effect of deep brain stimulation surgery on movement-related cortical potentials in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Patients who have had deep brain stimulation surgery for Parkinson's disease at Mayo Clinic Arizona will have electroencephalographic (EEG) measurements with the stimulator on followed by EEG measurements with the stimulator off. Patients who are scheduled to have deep brain stimulation surgery for Parkinson's disease will have EEG measurements before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had deep brain stimulation surgery for Parkinson's disease at Mayo Clinic Arizona, or who are scheduled to have deep brain stimulation surgery for Parkinson's disease at Mayo Clinic Arizona.

Exclusion Criteria:

* Patients unable to do repetitive dorsiflexion of the wrist due to orthopedic problems.
* Pregnant women.
* Prisoners or institutionalized individuals.

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary measures are six EEG bereitschaftspotential areas and amplitudes. | 12 months

SECONDARY OUTCOMES:
Unified Parkinson's disease rating scale score. | At time of EEG measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Evidente, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No